CLINICAL TRIAL: NCT06815380
Title: A European, Multicenter, Prospective Observational Phase IV Clinical Study to Assess the Impact of Lebrikizumab on Health-Related Well-Being and Control of Skin Manifestations in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study to Assess the Impact of Lebrikizumab on Health-Related Well-Being and Control of Skin Manifestations in Participants With Moderate-to-Severe Atopic Dermatitis
Acronym: ADTrust
Status: Recruiting | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: M-17923-35
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants: Participants with atopic dermatitis and treated with lebrikizumab (Ebglyss®) according to Summary of Product Characteristics (SmPC) in routine clinical practice, data will be collected and observed for 104 weeks.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is non-interventional study.

SUMMARY:
The main purpose of this study is to evaluate the impact of lebrikizumab treatment on the overall well-being of adult participants with moderate-to-severe AD in real-world clinical practice settings across Europe, as measured using validated 5-item World Health Organization Well-being Index (WHO-5) and to investigate effectiveness and safety of lebrikizumab, treatment satisfaction, and long-term effect of lebrikizumab treatment on participants in terms of disease symptomatology/control, fatigue, work impairment, patient's relationship with their skin, and overall QOL among adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult (greater than or equal to [>=] 18 years) male or female participants with diagnosis of moderate-to-severe Atopic dermatitis.
* Adult participants prescribed lebrikizumab as part of routine/usual care to manage their moderate-to severe Atopic dermatitis.
* Willingness and ability to participate in the study; participants must give their written consent to participate.

Exclusion Criteria:

* Hypersensitivity to the active substances or to any of the excipients of lebrikizumab (Ebglyss®).
* Participants with pre-existing helminth infections. These participants should be treated for helminth infection before starting lebrikizumab therapy.
* Concomitant use of live and live attenuated vaccines.
* Pregnant women, except when the potential benefit justifies the potential risk.
* Participants included in a clinical trial at baseline or at any time during the planned study period.
* Participants unable to comply with the requirements of the study or who, in the opinion of the study physician, should not participate in the study.
* Participants for whom medical chart is inaccessible to physicians to complete baseline data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderate to severe atopic dermatitis treated with lebrikizumab (Ebglyss®) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Absolute Measures in the Overall Health-related Well-being Index Evaluated Through World Health Organization (WHO-5) Score Throughout the Study Observation Period | Baseline up to Week 104
  The WHO-5 item well-being index is a generic global rating scale measuring subjective well-being and contains positively phrased items. The respondent is asked to rate how well each of the 5 items applies to him or her when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). The raw score therefore theoretically ranges from 0 (absence of well-being) to 25 (maximal well-being). To standardize the score on a scale from 0 (absent) to 100 (maximal), it is recommended to multiply the raw score by 4.
Change From Baseline in the Overall Health-related Well-being Index Evaluated Through WHO-5 Score Throughout the Study Observation Period | Baseline up to Week 104
  The WHO-5 item well-being index is a generic global rating scale measuring subjective well-being and contains positively phrased items. The respondent is asked to rate how well each of the 5 items applies to him or her when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). The raw score therefore theoretically ranges from 0 (absence of well-being) to 25 (maximal well-being). To standardize the score on a scale from 0 (absent) to 100 (maximal), it is recommended to multiply the raw score by 4.

SECONDARY OUTCOMES:
Percentage of Participants with 50 Percent (%) or Greater Reduction From Baseline in Overall Eczema Area and Severity Index (EASI) Score (EASI50) Throughout the Study Observation Period | Baseline up to Week 104
  The EASI is used to assess the severity and extent of AD; The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe). The EASI score was obtained by weight-averaging these 4 scores, resulting in the EASI score ranging from 0 to 72 where 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe, with higher values indicating more severe and or extensive disease. EASI 50 is defined as 50% or greater reduction from baseline in the EASI score.
Percentage of Participants with 75% or Greater Reduction From Baseline in Overall EASI Score (EASI75) Throughout the Study Observation Period | Baseline up to Week 104
  The EASI is used to assess the severity and extent of AD; The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe). The EASI score was obtained by weight-averaging these 4 scores, resulting in the EASI score ranging from 0 to 72 where 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe, with higher values indicating more severe and or extensive disease. EASI75 is defined as 75% or greater reduction from baseline in the EASI score.
Percentage of Participants with 90% or Greater Reduction From Baseline in Overall EASI Score (EASI90) Throughout the Study Observation Period | Baseline up to Week 104
  The EASI is used to assess the severity and extent of AD; The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe). The EASI score was obtained by weight-averaging these 4 scores, resulting in the EASI score ranging from 0 to 72 where 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe, with higher values indicating more severe and or extensive disease. EASI 90 is defined as 90% or greater reduction from baseline in the EASI score.
Percentage of Participants with 100% Reduction From Baseline in Overall EASI Score (EASI100) Throughout the Study Observation Period | Baseline up to Week 104
  The EASI is used to assess the severity and extent of AD; The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe). The EASI score was obtained by weight-averaging these 4 scores, resulting in the EASI score ranging from 0 to 72 where 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe, with higher values indicating more severe and or extensive disease. EASI100 is defined as 100% reduction from baseline in the EASI score.
Percentage of Participants With Absolute EASI Score Less than or Equal (<=) to 7 Throughout the Study Observation Period | Baseline up to Week 104
  The EASI is used to assess the severity and extent of AD; The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe). The EASI score was obtained by weight-averaging these 4 scores, resulting in the EASI score ranging from 0 to 72 where 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe, with higher values indicating more severe and or extensive disease.
Percentage of Participants with Overall Investigator Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) Throughout the Study Observation Period | Baseline up to Week 104
  The IGA is an instrument used to globally rate the severity of the participants AD. It is based on a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe), and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point. The score is based on an overall assessment of the degree of erythema, induration/papulation, lichenification, and oozing/crusting.
Absolute Measures in Overall IGA Score Throughout the Study Observation Period | Baseline up to Week 104
  The IGA is an instrument used to globally rate the severity of the participants AD. It is based on a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe), and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point. The score is based on an overall assessment of the degree of erythema, induration/papulation, lichenification, and oozing/crusting.
Change from Baseline in Overall IGA Score Throughout the Study Observation Period | Baseline up to Week 104
  The IGA is an instrument used to globally rate the severity of the participants AD. It is based on a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe), and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point. The score is based on an overall assessment of the degree of erythema, induration/papulation, lichenification, and oozing/crusting.
Absolute Measures in Patient-Oriented Eczema Measure (POEM) Score Throughout the Study Observation Period | Baseline up to Week 104
  The POEM is a 7-item, validated, questionnaire used by the participants to assess disease symptoms over the last week. The participants will be asked to respond to 7 questions on skin dryness, itching, flaking, cracking, sleep disturbance, bleeding and weeping. All 7 answers carry equal weight with a total possible score from 0 to 28 (answers scored as: No days=0; 1- 2 days = 1; 3-4 days = 2; 5-6 days = 3; everyday = 4). A high score is indicative of severe atopic dermatitis
Change From Baseline in POEM Score Throughout the Study Observation Period | Baseline up to Week 104
  The POEM is a 7-item, validated, questionnaire used by the participants to assess disease symptoms over the last week. The participants will be asked to respond to 7 questions on skin dryness, itching, flaking, cracking, sleep disturbance, bleeding and weeping. All 7 answers carry equal weight with a total possible score from 0 to 28 (answers scored as: No days=0; 1- 2 days = 1; 3-4 days = 2; 5-6 days = 3; everyday = 4). A high score is indicative of severe atopic dermatitis
Absolute Measures in Pruritus Numerical Rating Scale (NRS) Score Throughout the Study Observation Period | Baseline up to Week 104
  Pruritus NRS is a self-administered scale to assess participants worst level of itching on the skin (in the last 24 hours) experienced due to atopic dermatitis. The scale has a single-item that describes the worst level of itching on the skin due to atopic dermatitis in the last 24 hours on an 11-point scale anchored at 0 (no itching) and 10 (worst itching imaginable).
Change From Baseline in Pruritus NRS Score Throughout the Study Observation Period | Baseline up to Week 104
  Pruritus NRS is a self-administered scale to assess participants worst level of itching on the skin (in the last 24 hours) experienced due to atopic dermatitis. The scale has a single-item that describes the worst level of itching on the skin due to atopic dermatitis in the last 24 hours on an 11-point scale anchored at 0 (no itching) and 10 (worst itching imaginable).
Absolute Measures in Skin Pain NRS Score Throughout the Study Observation Period | Baseline up to Week 104
  Skin pain NRS is a self-administered scale to assess participants worst level of skin pain (in the last 24 hours) experienced due to atopic dermatitis. The scale has a single-item that describes the worst level of skin pain due to atopic dermatitis in the last 24 hours on an 11-point scale anchored at 0 (no skin pain) and 10 (worst skin pain imaginable).
Change From Baseline in Skin Pain NRS Score Throughout the Study Observation Period | Baseline up to Week 104
  Skin pain NRS is a self-administered scale to assess participants worst level of skin pain (in the last 24 hours) experienced due to atopic dermatitis. The scale has a single-item that describes the worst level of skin pain due to atopic dermatitis in the last 24 hours on an 11-point scale anchored at 0 (no skin pain) and 10 (worst skin pain imaginable).
Absolute Measures in Fatigue NRS Score Throughout the Study Observation Period | Baseline up to Week 104
  Fatigue NRS is a self-administered scale to assess participants worst level fatigue (in the last 24 hours) experienced due to atopic dermatitis. The scale has a single-item that describes the worst level of fatigue due to atopic dermatitis in the last 24 hours on an 11-point scale anchored at 0 (no fatigue) and 10 (worst fatigue imaginable).
Change From Baseline in Fatigue NRS Score Throughout the Study Observation Period | Baseline up to Week 104
  Fatigue NRS is a self-administered scale to assess participants worst level fatigue (in the last 24 hours) experienced due to atopic dermatitis. The scale has a single-item that describes the worst level of fatigue due to atopic dermatitis in the last 24 hours on an 11-point scale anchored at 0 (no fatigue) and 10 (worst fatigue imaginable).
Absolute Measures in Sleep Quality Scale Throughout the Study Observation Period | Baseline up to Week 104
  Sleep quality scale is a self-administered scale to assess participants overall sleep quality, in terms of the extent to which itching interfered with their sleep last night. The scale has a single-item that describes the interference of itching on sleep last night on an 11-point scale anchored at 0 (no interference) and 10 (unable to sleep at all).
Change From Baseline in Sleep Quality Scale Throughout the Study Observation Period | Baseline up to Week 104
  Sleep quality scale is a self-administered scale to assess participants overall sleep quality, in terms of the extent to which itching interfered with their sleep last night. The scale has a single-item that describes the interference of itching on sleep last night on an 11-point scale anchored at 0 (no interference) and 10 (unable to sleep at all).
Number of Participants With Adverse Events (AEs), Serious AEs, Adverse Drug Reactions (ADRs) and Serious ADRs Throughout the Study Observation Period | Baseline up to Week 104
  An AE is any untoward medical occurrence in a study participant who has been administered a medicinal product, and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. An ADR is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that there is a reasonable suspected causal relationship between the medicinal product and the adverse event. An AE or ADR is serious (SAE / SADR) as per following categories: death, is life-threatening, requires in-patient hospitalization or prolongs existing hospitalization, results in persistent or significant disability or incapacity, congenital anomaly or birth defect, or any other medically important event.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Augustin M, Bewley A, Bruggen MC, de Bruin-Weller MS, Ezzedine K, Ferrucci SM, Gkalpakiotis S, Herranz P, Johansson EK, Kampe T, Lapeere H, Legat FJ, Rehbinder EM, Szepietowski JC, Torres T, Vestergaard C, Werfel T, Domenech A, Massana E, Koscielny V, Narayanan S, Kasujee I, Gutermuth J. European, multicentre, prospective observational phase IV clinical study to assess the impact of lebrikizumab on health-related well-being and control of skin manifestations in patients with moderate-to-severe atopic dermatitis (ADTrust): study protocol. BMJ Open. 2025 Jul 11;15(7):e102155. doi: 10.1136/bmjopen-2025-102155. PMID 40645621